CLINICAL TRIAL: NCT03362294
Title: A Prospective, Multicenter, Two Arms, Open Label, Phase IIa Study to Assess the Safety and Efficacy of Once-a-month Long-acting Intramuscular Injection of 25 mg or 40mg Glatiramer Acetate (GA Depot) in Subjects With Primary Progressive Multiple Sclerosis (PPMS)
Brief Title: Safety and Efficacy of Monthly Long-acting IM Injection of 25mg or 40 mg GA Depot in Subjects With PPMS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mapi Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPMS-GA Depot 002
Record Dates: First submitted 2017-11-15; First posted 2017-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Primary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Intervention Model Description: The first 20 subjects are allocated to the 40mg arm and the last 10 subjects are allocated to the 25mg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GA Depot 40mg once monthly (Experimental): Monthly IM injection
  Interventions: Drug: GA Depot 40mg once monthly
- GA Depot 25mg once monthly (Experimental): Monthly IM injection
  Interventions: Drug: GA Depot 25mg once monthly

INTERVENTIONS:
Drug: GA Depot 40mg once monthly — Once-a-month long-acting intramuscular injection of 40mg Glatiramer Acetate (GA Depot)
  Arms: GA Depot 40mg once monthly
Drug: GA Depot 25mg once monthly — Once-a-month long-acting intramuscular injection of 25mg Glatiramer Acetate (GA Depot)
  Arms: GA Depot 25mg once monthly

SUMMARY:
This is a phase IIa study with GA Depot in subjects with Primary Progressive MS. GA Depot will be administered intramuscularly (IM), once every four weeks for 148 weeks.

The purpose of this study is to assess the safety and efficacy of GA Depot to slow the accumulation of disability progression in subjects with Primary Progressive MS.

DETAILED DESCRIPTION:
* 30 Subjects with a diagnosis of primary progressive multiple sclerosis (PPMS) who are not treated for PPMS at study entry (except for symptoms relief).
* Study product is GA long-acting injection (GA Depot) which is a combination of extended-release microspheres for injection and diluent (water for injection) for parenteral use. GA Depot will be administered intramuscularly (IM).
* The study duration for an individual subject in the core study will be 156 weeks, consisting of 4 weeks of screening evaluation (weeks -4 to 0), followed by a 148-week open-label treatment period, and a 4 weeks follow up period: through a total of 41 visits.
* Vital signs and safety assessment will be performed at each visit during the study.
* Physical examination will be performed at screening, baseline, 1 week after the second GA Depot treatment, 3 months after first GA Depot treatment and every 3 months thereafter. Last physical examination will be performed at FU visit.
* MRI will be performed at screenings and every 6 months thereafter until the end of the treatment period .
* Safety laboratory tests will be performed at screening, baseline, 1 month after first treatment, and every 3 months thereafter.
* Neurological assessment will be performed at screening, baseline, 3 months, and then every 3 months until end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects diagnosed with PPMS; Diagnosis of PPMS consistent with the McDonald Criteria (revisions of 2010).
2. Age between 18 and 65 years (inclusive).
3. Subjects diagnosed with PPMS for at least 1 year and with signs of disease progression in the year prior to screening, in a rate of ≥ 1 point increase / year in the EDSS score for EDSS between 2-5 and a rate of ≥0.5 point increase / year in the EDSS scores > 5.
4. EDSS ≥2 and ≤ 6.5 (Pyramidal or Cerebellar FS ≥ 2).
5. Documented history or the presence at screening of > 1 oligoclonal band (OCB) if quantitative testing was done, or OCB+ if not quantitative testing done and/or positive IgG index in the cerebrospinal fluid (CSF).
6. Women of child bearing potential must have a negative urine pregnancy test at screening and use an adequate contraceptive method throughout the study.
7. Ability to provide written informed consent.

Exclusion Criteria:

1. Subjects with RRMS, SPMS, or PRMS.
2. Subjects with a documented history of clinical relapse events.
3. Any relevant medical, surgical, or psychiatric condition, laboratory value, or concomitant medication which, in the opinion of the investigator, makes the subject unsuitable for study entry or potentially unable to complete all aspects of the study.
4. Contraindications or inability to successfully undergo magnetic resonance imaging (MRI) scanning.
5. Subjects diagnosed with any other than MS systemic autoimmune disease that may impact the CNS with MS like lesions such as Sarcoidosis, Sjögren's syndrome, Systemic Lupus Erythematosus (SLE), Lyme disease, APLA syndrome, etc.. Subjects with stable local/organ autoimmune disease such as psoriasis, Cutaneous Lupus erythematosus, thyroiditis (Hashimoto, grave) etc. may be considered eligible upon the PI's discretion.
6. Severe anemia (hemoglobin <10 g/dL).
7. Abnormal renal function (serum creatinine >1.5xULN or creatinine clearance <30 ml/min).
8. Abnormal liver function (transaminases >2xULN).
9. Pregnant or breast-feeding women.
10. Treatment with any kind of steroids during the last month prior to screening visit.
11. History of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a known hypersensitivity to any component of the study drug, e.g. glatiramer acetate (GA), polylactic-co-glycolic acid (PLGA), polyvinyl alcohol (PVA).
12. Known or suspected history of drug or alcohol abuse.
13. Known as positive for HIV, hepatitis, VDRL, or tuberculosis.
14. Active malignant disease of any kind. However, a patient, who had a malignant disease in the past, was treated and is currently disease - free for at least 7 years, may be considered eligible, upon the PI and sponsor's discretion.
15. Previous treatment with B-cell-targeting therapies (e.g. rituximab, ocrelizumab, atacicept, belimumab or ofatumumab) within 6 months prior to screening visit.
16. Previous treatment with cladribine within 2 years prior to screening visit
17. Previous treatment with azathioprine, mitoxantrone or methotrexate within 6 months prior to screening visit.
18. Previous treatment with lymphocyte-trafficking modifiers (e.g. natalizumab, fingolimod) within 6 months prior to screening visit. Subjects should have a total lymphocyte count within normal range.
19. Previous treatment with beta interferons, intravenous immunoglobulin, plasmapheresis within 2 months prior to screening visit.
20. Previous treatment with any glatiramer acetate therapy within 3 months prior to screening visit.
21. Uncontrolled diabetes.
22. Participation in an investigational study drug within 30 days prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety (Adverse Events and Injection Site Reactions) | 152 weeks
  Assessment of Adverse events (AEs) & Injection Sites Reactions (ISRs)

SECONDARY OUTCOMES:
Efficacy (Confirmed Disease Progression) | 148 weeks
  Time to onset of Confirmed Disease Progression (CDP) assessed by Expanded Disability Status Scale (EDSS). EDSS is a method of quantifying disability in people with MS. The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Efficacy (Whole brain volume change) | 148 weeks
  MRI assessment of percent of whole brain volume change.
Efficacy (Cortical volume change) | 148 weeks
  MRI assessment of percent of cortical volume change.

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Karni, MD, Principal Investigator — Coordinating PI
Locations (7):
- Israel (5):
  - Mapi Pharma Research site 09, Haifa
  - Mapi Pharma Research site 07, Jerusalem
  - Mapi Pharma Research site 08, Petah Tikva
  - Mapi Pharma Research site 06, Rehovot
  - Mapi Pharma Research site 01, Tel Aviv
- Moldova (2):
  - Mapi Pharma Research site 20, Chisinau
  - Mapi Pharma Research site 22, Chisinau

IPD SHARING:
Plan to Share IPD: No